CLINICAL TRIAL: NCT02287064
Title: An Open-label Trial of Intravenous Immune Globulin (IVIG)in Treating Spinocerebellar Ataxias
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA IVIG 2014
Record Dates: First submitted 2014-11-05; First posted 2014-11-10 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Spinocerebellar Ataxias
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Immunoglobulins, Intravenous

ARMS (1):
- Intravenous Immune Globulin (IVIG) (Experimental)
  Interventions: Drug: Intravenous Immune Globulin (IVIG)

INTERVENTIONS:
Drug: Intravenous Immune Globulin (IVIG) — IVIG will be infused over a course of five days in the form of GAMMAGARD LIQUID 10% solution, available from Baxter. For neurological and autoimmune diseases 2 grams per kilogram of body weight is implemented for three months over a five day course once a month.
  There is very limited reliable dose ranging data for IVIG in the treatment of any condition, and most dosing has been empiric. In our experience, we have empirically observed a more potent immunomodulatory effect from "induction dose" IVIG (2 g/kg) continued each month, than with the "booster dose" maintenance dose of 1gm/kg. Though there is no category one evidence to support this practice, neither is there such evidence to refute it. Additionally, results from previous trials of IVIG in SCAs show this dosage to be relatively safe and effective at this rate of infusion

SUMMARY:
The purpose of this study is to learn how Intravenous Immune Globulin (IVIG) will affect Spinocerebellar Ataxia (SCA) symptoms and how it will affect motor and nervous system function in participants Subtypes of SCA to be examined will include SCA types 1, 2, 3, 6, 10 and 11.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with SCA types 1, 2, 3, 6, 10, or 11, diagnosed by a movement disorder specialist.
* Age 18 years to 80 years.
* Able to ambulate with or without assistance for 30 feet.
* Women of child-bearing potential must use a reliable method of contraception and must provide a negative pregnancy test at entry into the study.
* Serum creatine kinase, complete metabolic panel, complete blood count, liver function tests, renal function tests, platelets and EKG do not reveal clinically significant abnormalities (results obtained from primary care physician and dated within the past 6 months or obtained at screening visit).
* Stable doses of all medications for 30 days prior to study entry and for the duration of the study.
* Diagnosis of peripheral neuropathy. See exclusion criteria 3 for specific types of peripheral neuropathy to be excluded.
* Throughout the study, all possible efforts will be made to maintain subject levels of activity, exercise or physical therapy.
* Subject permission (informed consent).

Exclusion Criteria:

* Any unstable illness that in the investigator's opinion precludes participation in this study.
* Use of any investigational product within the past 30 days.
* Presence of diabetes (as determined by blood glucose labs within the past 6 months), nutritional deficiency causing neuropathy (vitamin B1, 3, 6, and 12 or vitamin E), injuries, autoimmune disorders (HIV, lupus, pediatric Guillain-Barre syndrome, neurosarcoidosis, monoclonal gammopathy), tumors, infections (leprosy), exposures to toxins (alcohol, arsenic, mercury), thyroid disease or hereditary causes (cerebral amyloid angiopathy) known to result in the presence of peripheral neuropathy.
* Dementia or other psychiatric illness that prevents the subject from giving informed consent (MMSE less than 25).
* Legal incapacity or limited legal capacity.
* Presence of severe renal disease (estimated creatinine clearance <50 mL/min) or hepatic disease (as evidenced by labs reported within the past 6 months).
* Clinically significantly abnormal white blood cell count, hemoglobin or platelet count (as evidenced by labs reported within the past 6 months).
* Immunoglobulin A, Vitamin B (1, 3, 6, or 12), vitamin E or folate deficiencies (evidenced by screening lab evaluations).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Scale for the Assessment and Rating Ataxia (SARA) | Will be assesed at abseline, day 14, day28 and day 56.
  The primary outcomes will be the changes in the patient's SARA total score and frequency and severity of adverse events.

SECONDARY OUTCOMES:
clinician and patient global impression of improvement (CGI and PGI) | Will be assesed at abseline, day 14, day28 and day 56.
  Secondary outcome measures will include changes in the following scales between baseline and study endpoint: clinician and patient global impression of improvement (CGI and PGI); neurologic dysfunction as assessed by STAND scores; 9-hole peg test times.
Neurologic dysfunction as assessed by STAND scores | Will be assesed at abseline, day 14, day28 and day 56.
  Secondary outcome measures will include changes in the following scales between baseline and study endpoint: clinician and patient global impression of improvement (CGI and PGI); neurologic dysfunction as assessed by STAND scores; 9-hole peg test times.
9-hole peg test | Will be assesed at abseline, day 14, day28 and day 56.
  Secondary outcome measures will include changes in the following scales between baseline and study endpoint: clinician and patient global impression of improvement (CGI and PGI); neurologic dysfunction as assessed by STAND scores; 9-hole peg test times.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Zesiewicz, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States